CLINICAL TRIAL: NCT06662890
Title: Supersaturated Oxygen Therapy Using Radial Artery Access to Prevent Left Ventricular Remodeling After Anterior ST-segment Elevation Myocardial Infarction: a Randomized, Controlled Trial
Brief Title: Heart Attack Blood Oxygen Therapy Trial
Acronym: SSO2 Radial MI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: British Heart Foundation (Other); Zoll Medical Corporation (Industry); Robertson Centre for Biostatistics - University of Glasgow (Unknown)
Responsible Party: Principal Investigator, Colin Berry, Professor of Cardiology and Imaging, NHS National Waiting Times Centre Board
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23/CARD/34
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-10

CONDITIONS: Myocardial Infarct; Remodeling, Left Ventricle
Keywords: myocardial infarction; primary percutaneous coronary intervention; heart failure; adverse ventricular remodelling; biomarkers; coronary microvascular function; PREMS; PROMS
MeSH Terms: conditions — Myocardial Infarction; Ventricular Remodeling; Heart Failure | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Supersaturated oxygen therapy using radial artery access (Experimental): Supersaturated O2 (SSO2) therapy immediately following primary percutaneous coronary intervention using radial artery access in the cardiac catheter laboratory.
  Interventions: Other: Supersaturated oxygen
- Control group (Sham Comparator): Control (sham) procedure in addition to standard care
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Other: Supersaturated oxygen — Supersaturated O2 (SSO2) therapy immediately following primary percutaneous coronary intervention (PCI) using radial artery access in the cardiac catheter laboratory.
  https://www.zoll.com/products/supersaturated-oxygen-therapy
  Arms: Supersaturated oxygen therapy using radial artery access
Other: Sham (No Treatment) — Control (sham) procedure involving wrist manipulation in addition to standard care.
  Arms: Control group

SUMMARY:
'Heart attack', known as acute ST-segment elevation myocardial infarction, is a leading cause of heart failure and death. A lack of blood and oxygen damages the heart muscle potentially causing heart failure and premature death.

During the past 25 years, despite intensive research efforts, few, if any new medicines have been shown to prevent heart failure after a heart attack. New treatment approaches are needed.

The standard treatment for a heart attack is for a doctor to reopen the blocked blood vessel. The treatment is called primary percutaneous coronary intervention, or 'primary PCI'. The doctor places a thin plastic tube in a blood vessel in the wrist. The doctor then passes a longer thin tube via the wrist into the blocked heart artery. A small balloon is then used to open the blockage and a thin metal tube (stent) is placed inside the blood vessel to keep it open. The patient then returns to the ward.

Supersaturated oxygen therapy is designed to increase the blood oxygen level after the stent has been placed. The treatment lasts for one hour. The treatment is approved (CE-mark, FDA-approved) for patients presenting to doctors within 6 hours of symptoms onset. Supersaturated oxygen therapy is supported by results from two prior studies (AMIHOT, AMIHOT-II). Previously, the approach involved passing the plastic tubes via the femoral artery in the groin, limiting adoption. Since using the wrist is now standard care approach for heart attack treatment, our idea is to give supersaturated oxygen therapy via the wrist rather than the groin.

In this research study, we aim to assess the feasibility, safety and potential benefits of increasing blood oxygen content in patients who have been treated for a heart attack. The novel aspects of the study including giving the therapy via the wrist, the dummy procedure (sham/placebo), the randomized treatment assignment (coin-flip, play of chance), and the masking (blinding) of the patient participating in the study and the attending clinical staff, investigators and outcome assessors.

Patients who have been successfully treated for a heart attack will be invited to give informed consent at the end of the procedure. Fifty-six patients who have experienced a heart attack affecting the main area of the heart (anterior wall) will receive supersaturated therapy, or a dummy procedure, for one hour. The dummy procedure involves local anesthetic in the wrist and a pressure band as would normally be done.

The study also involves measuring small vessel function before and after the supersaturated oxygen / dummy procedure, a heart MRI scan at 2-5 days and again 3 months later, health questionnaires and blood samples to assess heart injury and to be stored for future research.

The study will provide information on safety, feasibility and preliminary insights into potential benefits to patients. The study will clarify whether a much larger study is warranted.

DETAILED DESCRIPTION:
This study is an academic, investigator-initiated clinical trial.

The design involves prospective enrolment of patients with a diagnosis of acute, anterior ST-segment elevation myocardial infarction (STEMI) presenting within 6 hours of symptom and undergoing primary PCI with radial artery acess. The protocol begins after standard, primary percutaneous coronary intervention (PCI). The timepoint for randomization (time zero) is at the end of successful primary PCI. Eligibility criteria include successful completion of primary PCI, defined as TIMI flow grade 2-3 in the left anterior descending coronary artery.

Given that the initial point of urgent/emergency care is in the catheter laboratory, the consent process will involve an initial witnessed verbal informed consent followed by randomization. This approach is in line with prior research in our hospital, contemporary evidence, feedback from experts with lived experience and international practice guidelines [PMID: 37622654 PMID: 32143733]. The Patient Information Sheet and Consent form will be provided to patients and carers on the ward after the angiogram. If the patient agrees to continue in the study then written informed consent will be obtained on the ward.

The study assessments will involve a blood sample, coronary angiography, coronary physiology, cardiovascular magnetic resonance (CMR) imaging scans, health status questionnaires, and electronic case record linkage. If the patient is eligible to participate and agrees to have electronic health record linkage follow-up but no other assessments or procedures, then consent will be invited for electronic health record follow-up only (no visits).

Informed consent will initially be obtained following arrival in the catheter laboratory. Blood samples would be obtained following arterial sheath insertion before PCI (since hemodilution due to the volume of radiographic contrast media may confound the analysis) study begins at the end of standard care primary PCI. Patients who fulfil the eligibility criteria and who have given written witnessed informed assent will be randomly assigned (2:1) to the intervention group or the control group.

Coronary microvascular function will be assessed in all patients at the end of the standard care primary PCI. The diagnostic guidewire should be positioned in the left anterior descending coronary artery using X-ray fluoroscopy. This will be repeated at the end of the intervention / control procedure.

Intervention group SSO2 therapy involves withdrawal of arterial blood, extra-corporeal hyper-oxygenation (ZOLL Circulation Inc console), and infusion of the hyper oxygenated blood into the PCI-treated left anterior descending coronary artery. The hyper oxygenated blood is returned using a standard catheter positioned in the left main coronary artery, via radial artery access. Therefore, temporary radial artery access using one or both radial arteries is needed for the one-hour duration of the SSO2 therapy in the cardiac catheter laboratory. Blinding measures will be implemented, including after returning to the coronary care unit until the end of the study.

Control group To minimize bias, patients assigned to the control group would follow the same schedule as if they were assigned to the intervention group. A control procedure will be undertaken. This procedure will mimic the actual procedure but without additional artery access i.e. no oxygen catheter therapy. The control procedure will involve conscious sedation, local anesthetic given in the usual way in the radial area, manual pressure, activation of the ZOLL Circulation Inc console (without the blood circuit), and then application of the radial closure device. The patient will be cared for by the clinical team in the usual way. The patient will remain blind to treatment group allocation, including after returning to the coronary care unit until the end of the study. Blinding to treatment group assignment will be prospectively documented.

Participants will be followed up with in person contacts up to 1-year post enrolment. Electronic health records may be checked without participant contact into the longer term.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Ischemic time ≤6 hours from symptom onset
3. Acute anterior ST-segment elevation myocardial infarction
4. Infarct-related left anterior descending coronary artery TIMI flow grade 2-3 at the end of PCI
5. Radial artery access
6. Partial pressure of oxygen (PaO2) >80 mmHg (10.7 kPa)

Exclusion Criteria:

1. Proximal coronary artery stenosis that restricts blood flow with the SSO2 catheter in place
2. Post-PCI non-stented dissection or perforation.
3. Moderate - severe heart valve stenosis, insufficiency, pericardial disease, or non-ischaemic cardiomyopathy
4. Known pregnancy.
5. Cardiogenic shock
6. Contra-indication to anticoagulation
7. Acute mechanical complication e.g., ventricular septal rupture, pseudoaneurysm, mitral regurgitation
8. Hemoglobin <10 g/dL
9. Major bleeding or major surgery within the past two months
10. Contra-indication to cardiovascular magnetic resonance (CMR) imaging e.g., severe claustrophobia, metallic foreign body.
11. Lack of witness verbal consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2038-11-01 (Estimated)

PRIMARY OUTCOMES:
N-terminal pro-B-type natriuretic peptide | 3 months from baseline
  N-terminal pro-B-type natriuretic peptide plasma concentration, within-subject change post-enrolment during follow-up.

SECONDARY OUTCOMES:
Coronary microvascular function | 2 hours from baseline
  Coronary microvascular function measured by bolus thermodilution
Infarct size | 2-5 days after enrolment
  Size of myocardial infarction (% left ventricular mass) measured by contrast-enhanced cardiovascular magnetic resonance (CMR) imaging
Microvascular obstruction | 2-5 days after enrolment
  Microvascular obstruction (% left ventricular mass) measured by contrast-enhanced cardiovascular magnetic resonance (CMR) imaging
Myocardial hemorrhage | 2-5 days after enrolment
  Incident myocardial hemorrhage detected by contrast-enhanced cardiovascular magnetic resonance (CMR) imaging
Left ventricular remodeling | 3 months from baseline
  Left ventricular remodeling revealed by left ventricular end-systolic volume index (ml/m2) measured by cardiovascular magnetic resonance (CMR) imaging
Myocardial blood flow | 3 months from baseline
  Global hyperemic blood flow (ml/min/g myocardium) in the anterior wall revealed by adenosine stress perfusion cardiovascular magnetic resonance (CMR) imaging.
Health-related quality of life | 12 months
  Patient reported outcome measure: EQ-5D-5L is a tool to measure health outcomes with five dimensions and five levels of problems each
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 12 months
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) has been qualified by the U.S. Food and Drug Administration as a Clinical Outcome Assessment.
Duke Activity Status Index | 12 months
  The Duke Activity Status Index (DASI) questionnaire is a valid measure of cardiopulmonary fitness.
Serious adverse events | 12 months
  Serious adverse events will be prospectively assessed. The primary criterion for safety monitoring is the incidence of major bleeding events.

CONTACTS AND LOCATIONS:
Locations (1):
- Golden Jubilee National Hospital, Clydebank, Dunbartonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Sharing of anonymized data based on sponsor approval.
Supporting Information: Study Protocol
Time Frame: To be confirmed
Access Criteria: Bone fide researchers, subject to sponsor approval
URL: https://www.gla.ac.uk/

REFERENCES:
- [Background] Stone GW, Martin JL, de Boer MJ, Margheri M, Bramucci E, Blankenship JC, Metzger DC, Gibbons RJ, Lindsay BS, Weiner BH, Lansky AJ, Krucoff MW, Fahy M, Boscardin WJ; AMIHOT-II Trial Investigators. Effect of supersaturated oxygen delivery on infarct size after percutaneous coronary intervention in acute myocardial infarction. Circ Cardiovasc Interv. 2009 Oct;2(5):366-75. doi: 10.1161/CIRCINTERVENTIONS.108.840066. Epub 2009 Sep 15. PMID 20031745
- [Background] Falah B, Kotinkaduwa LN, Schonning MJ, Redfors B, de Waha S, Granger CB, Maehara A, Eitel I, Thiele H, Stone GW. Microvascular Obstruction in Patients With Anterior STEMI Treated With Supersaturated Oxygen. J Soc Cardiovasc Angiogr Interv. 2024 Apr 6;3(5):101356. doi: 10.1016/j.jscai.2024.101356. eCollection 2024 May. PMID 39132455
- [Background] Chen S, David SW, Khan ZA, Metzger DC, Wasserman HS, Lotfi AS, Hanson ID, Dixon SR, LaLonde TA, Genereux P, Ozan MO, Maehara A, Stone GW. One-year outcomes of supersaturated oxygen therapy in acute anterior myocardial infarction: The IC-HOT study. Catheter Cardiovasc Interv. 2021 May 1;97(6):1120-1126. doi: 10.1002/ccd.29090. Epub 2020 Jul 10. PMID 32649037
- [Background] Shin D, Dai N, Wilburn P, Choi KH, Lee SH, Kim HK, Maehara A, Stone GW, Myung Lee J. Effect of Supersaturated Oxygen Therapy on Coronary Microcirculatory Function in Patients With Anterior STEMI. JACC Cardiovasc Interv. 2023 Oct 9;16(19):2469-2471. doi: 10.1016/j.jcin.2023.08.001. Epub 2023 Sep 6. No abstract available. PMID 37676228
- [Background] Carrick D, Haig C, Ahmed N, Carberry J, Yue May VT, McEntegart M, Petrie MC, Eteiba H, Lindsay M, Hood S, Watkins S, Davie A, Mahrous A, Mordi I, Ford I, Radjenovic A, Oldroyd KG, Berry C. Comparative Prognostic Utility of Indexes of Microvascular Function Alone or in Combination in Patients With an Acute ST-Segment-Elevation Myocardial Infarction. Circulation. 2016 Dec 6;134(23):1833-1847. doi: 10.1161/CIRCULATIONAHA.116.022603. Epub 2016 Nov 1. PMID 27803036
- [Background] Carrick D, Haig C, Ahmed N, McEntegart M, Petrie MC, Eteiba H, Hood S, Watkins S, Lindsay MM, Davie A, Mahrous A, Mordi I, Rauhalammi S, Sattar N, Welsh P, Radjenovic A, Ford I, Oldroyd KG, Berry C. Myocardial Hemorrhage After Acute Reperfused ST-Segment-Elevation Myocardial Infarction: Relation to Microvascular Obstruction and Prognostic Significance. Circ Cardiovasc Imaging. 2016 Jan;9(1):e004148. doi: 10.1161/CIRCIMAGING.115.004148. PMID 26763281
- [Derived] Joshi FR, Petty M, Ng YW, Elliott H, Anderson R, Gordon D, Hanna R, Sykes R, Leonard S, Morrow A, Tan D, Kamdar A, Perumal R, Creech JL, Kellman P, Welsh P, McConnachie A, Berry C. Supersaturated oxygen therapy using radial artery access to prevent left ventricular remodeling after anterior ST-segment elevation myocardial infarction: a randomized, controlled trial. Am Heart J Plus. 2025 May 28;55:100556. doi: 10.1016/j.ahjo.2025.100556. eCollection 2025 Jul. PMID 40510547